CLINICAL TRIAL: NCT03765892
Title: Study of the Academic and Professional Course of Narcoleptic Patients (NARCOSCOL-NARCOVITAE)
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0314
Record Dates: First submitted 2018-12-04; First posted 2018-12-05 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Narcolepsy
MeSH Terms: conditions — Narcolepsy | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Adult Case Group: Adults with type 1 narcolepsy according to the ICSD3
  Interventions: Other: Questionnaire (Adult)
- Adult Control Group: Parents, cousins and / or friends of included narcoleptic adult patients, at least 18 years old and not suffering from narcolepsy.
  Interventions: Other: Questionnaire (Adult)
- Children Case Group: Children with type 1 narcolepsy according to the OCSD3
  Interventions: Other: Questionnaire (Children)
- Children Control Group: Close friends and cousins of included narcoleptic children, minor and not suffering from narcolepsy.
  Interventions: Other: Questionnaire (Children)

INTERVENTIONS:
Other: Questionnaire (Adult) — Patients and case control will have to respond to the study questionnaire on the online entry platform to compare the distribution of socio-professional categories.
  Answering the questionnaires will take 45 minutes.
  Groups: Adult Case Group; Adult Control Group
Other: Questionnaire (Children) — Patients and case control will have to respond to the study questionnaire on the online entry platform to compare the proportion of subjects having repeated grades.
  Answering the questionnaires will take 45 minutes.
  Groups: Children Case Group; Children Control Group

SUMMARY:
Narcolepsy is a chronic, disabling, and rare sleep disorder (prevalence 1/2500) characterized by excessive daytime sleepiness and, in some patients, falls in muscle tone related to emotions (cataplexies). It often begins in childhood or in young adults. Symptoms of narcolepsy are responsible for an important handicap in everyday life, and are often misunderstood by the family and professional environment. In addition, many comorbidities are associated with narcolepsy, such as depression, anxiety, or obesity.

Few studies have investigated the impact of narcolepsy on patients' academic background, socio-professional integration, and quality of life.

Narcoleptic patients may experience more difficulties in their academic and professional path than non-narcoleptic people. These difficulties would be multifactorial (related to the disease itself, comorbidities, external factors ...).

As a better understanding of these determinants could help to inform patients and guide them in their choices, this study propose to establish a comprehensive inventory of educational and professional trajectories of narcoleptic patients in France in order assess the specificity of the difficulties encountered by the people concerned in their life course and to appreciate the attitude of the academic and professional circle with respect to the disease.

This category 3 study (according to the French law "Loi Jardé") is based on the case-control model and will be conducted in all National Reference and Competence Centers for Narcolepsy and Hypersomnia. It will include a population of adult and paediatric patients. It will answer questions about work and schooling in these patients.

ELIGIBILITY:
Inclusion Criteria:

The case group:

* Children (6 years <age <18 years) or adults with type 1 narcolepsy diagnosed on:
* a clinic in favor of narcolepsy: excessive daytime sleepiness lasting for more than 3 months.
* cataplexy and an positive multiple sleep latency test (mean sleep latency ≤ 8 min and ≥ 2 SOREM) or a hypocretin dosage in the CSF <110pg / L.
* Patients followed in one of the centers participating in the research.

The control group:

* At least one person close to the case (cousins, close friends ...).
* For adults: same sex as the case and if possible same age (+/- 5 years).
* For minors: same sex and if possible same age (+/- 2 years).
* Person not suffering from narcolepsy.

Exclusion Criteria:

The case group:

* Patients refusing to participate.
* Patients who do not speak the French language (incompatible with the reading, the comprehension and the filling of the questionnaires).
* Patients whose diagnosis of type 1 narcolepsy is not certain and / or has type 2 narcolepsy.
* Patients with narcolepsy symptomatic of another neurological disease.

The group controls:

* Person refusing to participate.
* Person who does not speak French (incompatible with reading, understanding and filling out questionnaires).
* The brothers and sisters of the case cannot be witnesses of the study.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will focus on pediatric and adult patients with type 1 narcolepsy and followed up in one of the participating rare disease reference or competence centers.
  Two control banks will be constituted:
  1. an "adult control" bank whose age is greater than 18 years: may be composed of the parents of included narcoleptic children or cousins and friends of included adult narcoleptic patients
  2. a bank " child control' whose age is less than 18 years: may be composed of friends and cousins of included narcoleptic children.
Sampling Method: Non-Probability Sample
Enrollment: 1605 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
For adult : distribution of professional situations | 45 minutes (time to answering the questionnaire)
  Distribution of professional situations in narcoleptic adult patients and related non-narcoleptic topics (employed, unemployed, student, retired, housewife/husband). (data collection form "professional situation").
For children : proportion of children who repeated a grade | 45 minutes (time to answering the questionnaire)
  Proportion of children who repeated a grade in narcoleptic children and non-narcoleptic control children ("school status" data collection form).

CONTACTS AND LOCATIONS:
Locations (18):
- France (18):
  - Centre de médecine du Sommeil CHU d'Angers, Angers
  - Service d'Explorations Fonctionnelles du Système Nerveux, Clinique du Sommeil, CHU de Bordeaux Groupe Hospitalier Pellegrin, Bordeaux
  - Unité de sommeil pédiatrique - Hôpital femme Mère Enfant - Hospices civils de Lyon, Bron
  - Service de neurophysiologie clinique CHU de Dijon, Dijon
  - Service de physiologie et Exploration fonctionnelle - Unité du Sommeil Hôpital Raymond Poincarré, Garches
  - Service de Neurophysiologie Clinique, Hôpital Roger Salengro, Lille
  - Centre de Médecine du Sommeil et des Maladies respiratoires - Centre Hospitalier de la Croix Rousse - Hospices Civils de Lyon, Lyon
  - Service de neurophysiologie clinique - centre du sommeil - Hôpital de la Timone, Marseille
  - Service de Neurologie - Troubles du Sommeil Hôpital Gui de Chauliac, Montpellier
  - Laboratoire d'Explorations Fonctionnelles Neurologiques, CHU de Nantes, Nantes
  - Centre du Sommeil et de la vigilance - Centre de référence Hypersomnies rares - Hôpital de l'Hôtel Dieu, Paris
  - Service de Physiologie Explorations fonctionnelles Hôpital Bichat Claude Bernard, Paris
  - Service des pathologies du sommeil Hôpital Pitié-Salpêtrière, Paris
  - Centre pédiatrique des pathologies du sommeil APHP CHU Robert Debré - Paris, Paris
  - Service de Neurophysiologie Clinique et Centre du Sommeil, CHU de Poitiers, Poitiers
  - Centre des Troubles du Sommeil, Hospices Civils de Strasbourg, Strasbourg
  - Explorations Neurophysiologiques, Hôpital Pierre Paul Riquet, CHU Toulouse Purpan, Toulouse
  - Centre du Sommeil du Service de Neurologie et de Neurophysiologie Clinique - CHRU Bretonneau, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peter-Derex L, Fort E, Putois B, Martel N, Ricordeau F, Bastuji H, Arnulf I, Barateau L, Bourgin P, Dauvilliers Y, Debs R, Dodet P, Dudoignon B, Franco P, Hartley S, Lambert I, Lecendreux M, Leclair-Visonneau L, Leger D, Lemesle-Martin M, Leotard A, Leu-Semenescu S, Limousin N, Lopez R, Meslier N, Micoulaud-Franchi JA, Charley-Mocana C, d'Ortho MP, Philip P, Ruppert E, de La Tullaye S, Brigandet M, Margier J, Rolland B, Charbotel B, Mazza S. Effort/reward imbalance and comorbidities burden in academic and professional careers of patients with narcolepsy type 1. J Clin Sleep Med. 2025 Jun 1;21(6):983-997. doi: 10.5664/jcsm.11598. PMID 39943847